CLINICAL TRIAL: NCT04021342
Title: The Effect of Tart Cherry (Prunus Cerasus) Concentrate on Cardiometabolic Risk Factors, Exercise Capacity and Cognitive Function
Brief Title: The Effect of Tart Cherry (Prunus Cerasus) Concentrate on Physiological and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Cherry Marketing Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4240
Record Dates: First submitted 2019-05-29; First posted 2019-07-16 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cardiometabolic Risk Factors; Cognitive Function; Exercise Capacity
Keywords: Tart cherry; Montmorency cherries; Prunus Cerasus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The treatment drink (tart cherry concentrate) and placebo are matched for colour and packed in identical plastic containers. The assigned beverages are packed and given to the participants by an independent researcher not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montmorency tart cherry concentrate (Active Comparator): Participants will consume 30 ml of Montmorency tart cherry concentrate (MC) concentrate (King Orchard farms, USA) twice daily, once in the morning and again in the evening. According to the manufacturer each 30 ml dose of MC is estimated to be equivalent to approximately 90 whole cherries (equating to ~180 cherries per day).
  Interventions: Dietary Supplement: Montmorency tart cherry concentrate
- Isocaloric cherry flavoured placebo (Placebo Comparator): The PLA is prepared by mixing by mixing unsweetened black cherry flavoured Kool-Aid (Kraft Foods, United States), dextrose, fructose with water to best match the calorie content of the MC concentrate. Additional lemon juice, for tartness, and artificial food colouring is added so the final product had a similar visual properties to the active comparator.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Montmorency tart cherry concentrate — Based on previous analysis done by our laboratory each 60 ml of Montmorency tart cherry concentrate contains approximately 73.5 mg of anthocyanins (cyanidin-3-glucoside equivalents) and 178.8 mg of total phenolics (mean gallic acid equivalents)
  Arms: Montmorency tart cherry concentrate
Dietary Supplement: Placebo — Placebo beverage matched for calorie content and visual properties of the cherry concentrate
  Arms: Isocaloric cherry flavoured placebo

SUMMARY:
A randomized, double blind, counterbalanced, placebo controlled independent groups design to determine the effects of 3 month supplementation with tart cherry concentrate on indices of cardiometabolic health, exercise capacity and cognitive function. Following screening and recruitment, participants are familiarised with the testing equipment and procedures after which they will be randomly assigned to receive either Montmorency tart cherry concentrate (MC) or an isocaloric placebo (PLA), stratified by gender. The study is comprised of two experimental visits and outcome variables are assessed at baseline (before supplementation) and at 3 months (follow up; after supplementation).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 40-60 years
* consume on average ≤5 servings of fruits and vegetables per day
* additionally have ≥1 risk factor for type 2 diabetes

Exclusion Criteria:

* not regularly taking medication (or stabilised ≥ 3 months, with no adverse symptoms) or antioxidant supplements
* history of cardiometabolic, gastointestinal disease or malabsorption syndromes
* stage 2 hypertension (SBP >159 mm Hg or DBP >99 mm Hg)
* individuals who report changes in dietary or physical activity patterns within 3 months
* vegetarians, vegans or known eating disorders
* alcohol intake of more than 21 units per week
* BMI ≥40 kg/m2
* are pregnant or planning to become pregnant during the study, lactating, or initiating or changing a hormone replacement therapy regimen within 3 months of the start of the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Change from baseline at 3 months
  Systolic blood pressure (mmHg) Diastolic blood pressure (mmHg)
Arterial Stiffness | Change from baseline at 3 months
  Pulse wave velocity (m/s)
Arterial Stiffness | Change from baseline at 3 months
  Augmentation index (%)
Endothelial function | Change from baseline at 3 months
  Flow mediated dilation (% change)

SECONDARY OUTCOMES:
Indices of metabolic health | Change from baseline at 3 months
  glucose (mmol/L) triglycerides (mmol/L) LDL cholesterol (mmol/L) HDL cholesterol (mmol/L)
Cognitive function | Change from baseline at 3 months
  Computerized cognitive function assessment percentage accuracy (%)
Cognitive function | Change from baseline at 3 months
  Computerized cognitive function assessment reaction time (m/s)
Cerebral Blood flow | Change from baseline at 3 months
  Oxygenated heamoglobin (Oxyhb)
Cerebral Blood flow | Change from baseline at 3 months
  Deoxygenated heamoglobin (deoxyhb)
Exercise Capacity | Change from baseline at 3 months
  Estimated aerobic exercise capacity (VO2max) measured by a submaximal cycling test

OTHER OUTCOMES:
Body composition | Change from baseline at 3 months
  Fat mass (g) Lean mass (g)
Body composition | Change from baseline at 3 months
  Fat percentage (%)
Body composition | Change from baseline at 3 months
  Android/gynoid ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No